CLINICAL TRIAL: NCT03349463
Title: Evaluation of Fluciclovine Uptake in Patients With Cervical, Ovarian Epithelial or Endometrial Cancers. Pilot Study.
Brief Title: Evaluation of Fluciclovine Uptake in Patients With Cervical, Ovarian Epithelial or Endometrial Cancers.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bital Savir-Baruch (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor-Investigator, Bital Savir-Baruch, Nuclear Medicine Assistant Professor, Loyola University
Organization: Loyola University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 209877
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Cervical Cancer; Endometrial Cancer; Ovarian Epithelial Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Carcinoma, Ovarian Epithelial | interventions — fluciclovine F-18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- 18F-Fluciclovine (Experimental)
  Interventions: Drug: Fluciclovine F18

INTERVENTIONS:
Drug: Fluciclovine F18 — All study participants will receive 10 mCi of 18F-Fluciclovine (Axumin) one time administered through injection through the catheter into participant's arm immediately before PET/CT scan.
  Other Names: Axumin; anti-3-[18F] FACBC

SUMMARY:
An important part of staging and deciding the method of treatment is knowing areas of how cancer is involved. Diagnostic imaging is often used to determine the location of the cancer using techniques like nuclear medicine, MRI (magnetic resonance imaging), CT (computerized tomography), and ultrasound. Each technique looks for cancer in different ways and are often used together to make a better determination of the extent of disease.

One of the techniques used in cancer imaging is PET/CT. This technique combines a nuclear medicine study (PET or positron emission tomography) with CT performing both scans at the same time. PET/CT most commonly uses a radioactive sugar (FDG or fluorodeoxyglucose) to detect the cancer. The problem with FDG is that it is excreted by the kidneys and collected in the bladder. Even though the bladder is emptied prior to the scan, the FDG activity present there may interfere with the detection of small areas of cancer involvement in lymph nodes or adjacent areas. It is because of this that PET/CT using FDG is infrequently used in gynecological cancers.

This purpose of this study is to evaluate if 18F-fluciclovine can be used to help determine the extent of gynecological cancers. 18F-fluciclovine (also known as AXUMIN) is a radioactive tracer which has been approved by the FDAFood and Drug Administration (FDA) for use in patients with prostate cancer. 18F-fluciclovine has much less excretion through the kidneys which improves the PET/CT imaging of the pelvis.

ELIGIBILITY:
Inclusion Criteria:

* GYN cancer (ovarian, endometrial, or cervical) was biopsy-proven and/or schedule for subsequent surgery based on clinical presentation (imaging, markers)
* Age ≥ 18 years.
* Can tolerate 18F-fluciclovine PET/CT exam (can lie on her back for the duration of the scan).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Ongoing systemic therapy for cancer
* Systemic therapy for cancer in the past 3 months
* Inability to tolerate 18F-fluciclovine PET/CT exam
* Pregnant or lactating women

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
18F-Fluciclovine uptake in gynecologic neoplasms | Day 30
  PET/CT imaging

CONTACTS AND LOCATIONS:
Overall Officials: Bital Savir-Baruch, M.D, Principal Investigator — Nuclear Medicine Assistant Professor
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Atri M, Zhang Z, Dehdashti F, Lee SI, Ali S, Marques H, Koh WJ, Moore K, Landrum L, Kim JW, DiSilvestro P, Eisenhauer E, Schnell F, Gold M. Utility of PET-CT to evaluate retroperitoneal lymph node metastasis in advanced cervical cancer: Results of ACRIN6671/GOG0233 trial. Gynecol Oncol. 2016 Sep;142(3):413-9. doi: 10.1016/j.ygyno.2016.05.002. Epub 2016 Jul 27. PMID 27178725
- [Background] Cannistra SA. Cancer of the ovary. N Engl J Med. 2004 Dec 9;351(24):2519-29. doi: 10.1056/NEJMra041842. No abstract available. PMID 15590954
- [Background] Khiewvan B, Torigian DA, Emamzadehfard S, Paydary K, Salavati A, Houshmand S, Shamchi SP, Werner TJ, Aydin A, Roy SG, Alavi A, Kumar R. Update of the role of PET/CT and PET/MRI in the management of patients with cervical cancer. Hell J Nucl Med. 2016 Sep-Dec;19(3):254-268. doi: 10.1967/s002449910409. Epub 2016 Nov 8. PMID 27824966
- [Background] Kim TH, Kim J, Kang YK, Lee M, Kim HS, Cheon GJ, Chung HH. Identification of Metabolic Biomarkers Using Serial 18F-FDG PET/CT for Prediction of Recurrence in Advanced Epithelial Ovarian Cancer. Transl Oncol. 2017 Jun;10(3):297-303. doi: 10.1016/j.tranon.2017.02.001. Epub 2017 Mar 15. PMID 28314183
- [Background] Kizer NT, Zighelboim I, Case AS, Dewdney SB, Thaker PH, Massad LS. The role of PET/CT in the management of patients with cervical cancer: practice patterns of the members of the Society of Gynecologic Oncologists. Gynecol Oncol. 2009 Aug;114(2):310-4. doi: 10.1016/j.ygyno.2009.04.018. Epub 2009 May 14. PMID 19446317
- [Background] Rockall AG, Cross S, Flanagan S, Moore E, Avril N. The role of FDG-PET/CT in gynaecological cancers. Cancer Imaging. 2012 Mar 5;12(1):49-65. doi: 10.1102/1470-7330.2012.0007. PMID 22391444
- [Background] Signorelli M, Guerra L, Buda A, Picchio M, Mangili G, Dell'Anna T, Sironi S, Messa C. Role of the integrated FDG PET/CT in the surgical management of patients with high risk clinical early stage endometrial cancer: detection of pelvic nodal metastases. Gynecol Oncol. 2009 Nov;115(2):231-5. doi: 10.1016/j.ygyno.2009.07.020. Epub 2009 Aug 19. PMID 19695685
- [Background] Jager PL, Vaalburg W, Pruim J, de Vries EG, Langen KJ, Piers DA. Radiolabeled amino acids: basic aspects and clinical applications in oncology. J Nucl Med. 2001 Mar;42(3):432-45. PMID 11337520
- [Background] Washburn LC, Sun TT, Anon JB, Hayes RL. Effect of structure on tumor specificity of alicyclic alpha-amino acids. Cancer Res. 1978 Aug;38(8):2271-3. PMID 208763
- [Background] Washburn LC, Sun TT, Byrd B, Hayes RL, Butler TA. 1-aminocyclobutane[11C]carboxylic acid, a potential tumor-seeking agent. J Nucl Med. 1979 Oct;20(10):1055-61. PMID 231642
- [Derived] Savir-Baruch B, Lovrec P, Solanki AA, Adams WH, Yonover PM, Gupta G, Schuster DM. Fluorine-18-Labeled Fluciclovine PET/CT in Clinical Practice: Factors Affecting the Rate of Detection of Recurrent Prostate Cancer. AJR Am J Roentgenol. 2019 Oct;213(4):851-858. doi: 10.2214/AJR.19.21153. Epub 2019 Jun 19. PMID 31216198